CLINICAL TRIAL: NCT03122171
Title: Use of Low Cost Prostheses to Improve Upper Extremity Function in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-02093
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Palsy; Prosthesis User
MeSH Terms: conditions — Cerebral Palsy | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prosthesis (Experimental)
  Interventions: Other: Occupational Therapy Treatment

INTERVENTIONS:
Other: Occupational Therapy Treatment — Each occupational therapy treatment will be a one-hour standardized session that will include the following: stretching/strengthening (approximately 20 minutes), bi-manual training (approximately 20 minutes), and activities of daily living (approximately 20 minutes).

SUMMARY:
The purpose of the study is to assess the effectiveness of an upper extremity prosthesis in improving the upper extremity function of children with cerebral palsy who have limited use of their hands. Twelve children, aged 4-17 years, who have cerebral palsy and limitations in their ability to use their hands, will be enrolled. All participants will be fitted with a 3D printed arm/hand prosthesis and receive 8 occupational therapy sessions. Each subject will be evaluated pre-treatment, post-occupational therapy sessions and at 6 months follow-up. The evaluation will include assessment of (1)passive and active arm/hand movement and (2)functional hand skills using several standardized tests. The results from the pre-treatment and the two post-treatment evaluations will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: cerebral palsy
* 4-17 years old
* MACS levels III - V
* Active movement of wrist or elbow

Exclusion Criteria:

* MACS levels I, II
* Botox or orthopedic surgery in past 6 months
* Severe contractures
* Lack of voluntary arm motion

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Chu, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prosthesis
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prosthesis
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 15.8 [13 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Increase in Assisting Hand Assessment (AHA) Score
Description: The Assisting Hand Assessment (AHA) is a test of hand function in children with difficulties using one of their hands. The AHA measures how effectively the affected hand and arm is used in bimanual performance. An assessment is performed by observing the child's spontaneous handling of toys in a relaxed and playful session. Scores based on 22-items on a 4-point rating scale evaluating quality of the performance (1=does not do, 4=effective). The range of sum scores is 22-88 points. A clinical significant increase in score indicates an increase in quality of performance.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
Participants | 4

2. Primary Outcome: Number of Participants With Increase in Pediatric Motor Ability Log (PMAL) Scores Post-Treatment
Description: The PMAL is a structured interview in which the caregiver reports "How Often" (amount) and "How Well" (quality of movement) the child uses their involved upper limb when completing 22 activities of daily living. Scores range from 0-10; the higher the score, the better the quality of movement. An increase in PMAL score indicates a higher amount of upper extremity use and better quality of movement.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
Participants | 4

3. Primary Outcome: Number of Participants With Increase in Melbourne Assessment 2 (MA2) Scores
Description: The Melbourne Assessment 2 (MA2) is a valid and reliable criterion-referenced test for evaluating four elements of upper limb movement quality in children with a neurological impairment aged 2.5 to 15 years: (i) Range of motion, (ii) Accuracy of reach and placement, (iii) Dexterity of grasp, release and manipulation and (iv) Fluency of movement. An increase in score indicates an increase in upper limb movement quality.
Time Frame: Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
Participants
  Range of Motion | 4
  Accuracy of Reach and Placement | 3
  Dexterity of Grasp | 3
  Fluency of Movement | 2

4. Secondary Outcome: Number of Participants With Increase in Pediatric Quality of Life Inventory Subtest Scores Post-Treatment
Description: The PedsQL is a brief, standardized, generic assessment instrument that systematically assesses patients' and parents' perceptions of HRQOL in pediatric patients with chronic health conditions using pediatric cancer as an exemplary model. 7 sub-tests will be reported on. Higher scores indicate better HRQOL (Health-Related Quality of Life), an increase in score indicates an increase in HRQOL.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
Participants
  Daily Activities | 3
  School Activities | 3
  Movement and Balance | 3
  Pain and Hurt | 2
  Fatigue | 1
  Eating Activities | 1
  Speech and Communication | 1

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03122171/Prot_000.pdf